CLINICAL TRIAL: NCT06341322
Title: Using Behavioural and Cultural Insights to Understand and Address Barriers and Drivers to Colorectal Cancer Home-testing in Croatia
Brief Title: Using Behavioural and Cultural Insights to Increase Colorectal Cancer Home-testing in Croatia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Veerle Snijders (Other)
Collaborators: Croatian Institute of Public Health (Unknown); Andrija Štampar School of Public Health (Unknown)
Responsible Party: Sponsor-Investigator, Veerle Snijders, Behavioural Scientist, World Health Organization
Organization: World Health Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: ERC0003996
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Behavior Change
Keywords: colorectal cancer; cancer screening; behavioral insights; communications
MeSH Terms: conditions — Colorectal Neoplasms; Communication

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either control (no reminder screening invitation) or one of three treatments (standard reminder letter, behaviorally informed reminder letter, behaviorally informed letter with home testing kit included).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants do not receive a reminder letter, which is treatment as usual.
- Standard letter (Experimental): Participants receive a reminder letter which is based on the current colorectal cancer screening invitation.
  Interventions: Behavioral: Standard letter
- Behaviorally informed letter (Experimental): Participants receive a reminder letter which incorporates several behavioral components, including an active choice prompt, social norm, simplification, chunking and call to action.
  Interventions: Behavioral: Behaviorally informed letter
- Behaviorally informed letter + testing kit (Experimental): Participants receive the behaviorally informed letter plus the colorectal home testing kit, which removes the current barrier of having to request a kit.
  Interventions: Behavioral: Behaviorally informed letter; Behavioral: Home testing colorectal cancer kit

INTERVENTIONS:
Behavioral: Standard letter — A reminder letter to encourage recipients to order the colorectal cancer home testing kit, based on the current invite letter.
  Arms: Standard letter
Behavioral: Behaviorally informed letter — A reminder letter to encourage recipients to order the colorectal cancer home testing kit, with incorporates severally behaviorally informed components, including an active choice prompt, social norm, call to action, chunking and simplification.
  Arms: Behaviorally informed letter; Behaviorally informed letter + testing kit
Behavioral: Home testing colorectal cancer kit — The home testing kit is included with the reminder letter, instead of the usual process of responding to the letter to order the kit
  Arms: Behaviorally informed letter + testing kit

SUMMARY:
Colorectal cancer (CRC) is one of the leading causes of death in Croatia. An average of 3600 cases are diagnosed and an average of 2100 people die from the disease every year. Since 2007, Croatia has invited every man and woman aged 50-74 to participate in the home testing screening programme every two years. Currently only around 36% of the invited request the test-kit and 25% complete the home testing procedure, far below the target of 40-60%.

The Croatian Institute of Public Health with technical support from World Health Organization (WHO) Regional Office for Europe is undertaking a mixed-methods research study with the aim to increase the completion of colorectal cancer home testing and improve our knowledge of the barriers and drivers to do so. The study has a quantitative and a qualitative component:

1. Quantitative: testing the introduction of a reminder letter to encourage people to respond to the initial invite to participate in the CRC home test program and test which elements of a reminder letter improve response rates.

   The quantitative component consists of a four-arm reminder letter randomized controlled trial (RCT) comparing no letter, standard letter, behaviorally informed letter, and behaviorally informed letter sent with a home testing kit to investigate the effectiveness of reminders in increasing uptake of home-testing for colorectal cancer. Recruitment and data collection for the reminder letter trial will be conducted utilizing the routine screening process and routinely collected screening data.
2. Qualitative: conducting in-depth interviews with people from the target population who did or did not respond to the CRC invite letter and reminder to better understand the barriers and drivers to participation.

The qualitative component consists of 24 in-depth interviews (IDIs) conducted with members of the target population to identify barriers and drivers to completing colorectal cancer screening home-testing. Data collection for IDIs will be face-to-face, using discussion guides, and will be audio recorded. The audio-recordings will then be analyzed using a rapid analysis approach based on by the modified Capability-Opportunity-Motivation-Behavior (COM-B) framework.

ELIGIBILITY:
Inclusion Criteria:

* eligible to participate in the national colorectal cancer screening programme
* live in a study location (Split-Dalmatia or Zagreb City counties)
* did not respond to the cancer screening invite letter

Exclusion Criteria:

* participated in the colorectal screening programme in the last 24 months

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13000 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Home test kit ordered | 5 weeks
  Did the participant order the colorectal cancer home testing kit? Routinely collected data.
Completed colorectal cancer screening | 5 weeks
  Did the participant complete the home testing kit and return it to the health authority? Routinely collected data.

SECONDARY OUTCOMES:
Opted out | 5 weeks
  Did the participant actively opt out of participating in the screening program? Routinely collected data.
Qualitative feedback | 10 weeks
  Qualitative feedback on the intervention arms and colorectal cancer screening experience. Collected through 24 semi-structured interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Croatian Institute of Public Health, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No
The study utilizes the data that is routinely collected as part the Croatian National Screening Database, only specific approved members of the screening program are able to access and utilize this data. For this reason, it is currently not planned to share individual participant data.